CLINICAL TRIAL: NCT03123289
Title: Novel Gallium 68 Citrate in Orthopedic Infections
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left the institute and the funding expired.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Nasrin Ghesani, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20160000134
Record Dates: First submitted 2017-04-04; First posted 2017-04-21 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Joint Prosthesis
Keywords: PET/CT; 68Gallium Citrate; Orthopedic Hardware infection

STUDY DESIGN:
Intervention Model Description: Same patients are scanned with two radiotracers within 24-48 hours. Results of the two scans are compared against each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 68Gallium-citrate (Experimental): This arm, undergoing the "68-Gallium citrate PET/CT scan intervention", includes the PET/CT scans performed with 68Gallium-citrate radiotracer. Note that same patients scanned with different radiotracers serve in both arms.
  Interventions: Drug: 68-Gallium citrate PET/CT scan
- 18F-FDG (Experimental): This arm, undergoing the "18F FDG PET/CT scan intervention", includes the PET/CT scans performed with 18F-FDG tracer.
  Note that same patients scanned with different radiotracers serve in both arms.
  Interventions: Drug: 18F FDG PET/CT scan

INTERVENTIONS:
Drug: 68-Gallium citrate PET/CT scan — After establishment of an intravenous access, approximately 5 mCi of 68Ga-citrate (Zevacor Molecular, Somerset, NJ, USA) will be administered intravenously. Whole body PET/CT scan will be performed after 60 minutes of uptake phase.
  Arms: 68Gallium-citrate
Drug: 18F FDG PET/CT scan — Subjects will undergo FDG PET/CT scan using the same imaging parameters either on the same day or within the next 24-48 hours. The subjects will be requested to fast for a minimum of 4 h prior to PET acquisition. After confirmation of a blood glucose level ≤200 mg/dl, technologists will establish the intravenous access and the subject will receive approximately 10 mCi of 18F-FDG (Zevacor Molecular, Somerset, NJ, USA) intravenously. The subject will be placed in uptake room for 60 minutes to allow for optimal localization of the compound. The subjects will be requested to void prior to administration of 18FDG and again prior to image acquisition.
  Arms: 18F-FDG

SUMMARY:
In the proposed study, our aim is to evaluate the uptake of 68Gallium-citrate in patients with failed joint prosthesis and compare it with that of conventional 18fluorine-fluorodeoxyglucose (18F-FDG) positron emission tomography/computed tomography (PET/CT) scan. We will perform PET/CT scan with 68Gallium citrate and 18F-FDG in subjects with failed hip or knee prosthesis. Both 68Gallium-citrate and 18F-FDG scans, done within 24-48 hours from each other, will be performed within 4 weeks before surgical evaluation/revision of the hardware.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months after hip replacement with complaint of joint pain.
* Radiographic studies compatible with prosthesis loosening (i.e. periprosthetic infection or aseptic loosening).
* Pending surgical evaluation and tissue sampling within the next few weeks to differentiate between infection and aseptic loosening.

Exclusion Criteria:

* Inability to consent
* Pregnancy or known or suspected hypersensitivity to metals or gallium
* Joint replacement for any reason other than primary or secondary osteoarthritis
* Prior surgical therapy for prosthesis failure after initial hospital discharge
* Active inflammatory/infectious process at any location other than prosthetic joint (Sarcoidosis, Rheumatoid arthritis, HIV infection, SLE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
68Gallium-citrate and 18F-FDG uptake (SUV) surrounding the femoral and acetabular components of the prosthesis | 1 year
  The radiotracer uptake in SUV units is measured in different Gruen zones around the prosthesis and normalized by that of the liver. The values of the two scans will be compared against each other for all patients.

SECONDARY OUTCOMES:
Sensitivity, specificity, and accuracy of 68Gallium-citrate and 18F-FDG scans, by using surgical pathology results as the gold standard. | 1 year
  Using the surgical histology and tissue culture as the gold standard, sensitivity and specificity of both techniques will be calculated. The aim is determine which modality has more accuracy to differentiate septic prosthesis failure from aseptic entities.

CONTACTS AND LOCATIONS:
Overall Officials: Nasrin Ghesani, MD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03123289/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03123289/SAP_001.pdf
  • Informed Consent Form (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03123289/ICF_002.pdf